CLINICAL TRIAL: NCT07349407
Title: The Effect of Dilute Epinephrine Saline Irrigation on Field Clarity in Ankle Arthroscopic Surgery Compared to a Tourniquet: a Double-blind, Randomized Controlled Trial
Brief Title: Dilute Epinephrine vs Tourniquet for Visualization in Ankle Arthroscopy: A RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-1632
Record Dates: First submitted 2025-12-21; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Chronic Ankle Instability; Ankle Ligament Injury; Ankle Arthroscopy
Keywords: Arthroscopic visual field

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study was conducted using a double-blind design. After concealed randomization, only the principal investigator had access to group assignments, while participants, observers, and surgeons were blinded and identified solely by subject numbers.
  Upon enrollment and signing of informed consent, participants were informed that they would be randomly assigned to either the epinephrine group or the tourniquet group. Observers received only the corresponding subject numbers from the principal investigator and were responsible for data collection and recording without knowledge of group allocation.
  For surgeons, both groups had an inflatable tourniquet placed at the standard position prior to surgery. After verification by all three parties (participant, investigator, and surgical team), the surgeon left the room for 15 minutes. Group-specific interventions (inflating the tourniquet or not) were implemented after surgical draping was completed. Surgeons were then called in to perform th
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epinephrine group (Experimental)
  Interventions: Drug: Epinephrine group
- Tourniquet group (Active Comparator)
  Interventions: Device: Tourniquet group

INTERVENTIONS:
Drug: Epinephrine group — Irrigation fluid consisted of normal saline mixed with 1 mL of 1:1000 epinephrine per 3-liter bag. A tourniquet was placed but left deflated as a rescue measure and could be inflated intraoperatively if necessary.
  Arms: Epinephrine group
Device: Tourniquet group — Standard tourniquet application
  Arms: Tourniquet group

SUMMARY:
This multicenter, prospective randomized controlled trial investigates the effect of dilute epinephrine irrigation versus tourniquet use on visual field clarity (VFC) during ankle arthroscopy. Patients are randomized into an epinephrine group (normal saline with 1 mL of 1:1000 epinephrine per 3 L bag; tourniquet placed but not inflated unless needed) or a standard tourniquet group. The primary outcome is arthroscopic visual field clarity assessed using a 4-point Likert-style numeric rating scale. Secondary outcomes include postoperative pain intensity at 2 and 24 hours (VAS), and the incidence of hypotension, bradycardia, and cardiovascular adverse events.

DETAILED DESCRIPTION:
Study Objective and Design

This study aims to evaluate the effect of dilute epinephrine irrigation versus tourniquet use on visual field clarity (VFC) during ankle arthroscopic surgery, while also assessing the incidence of hypotension/bradycardia events and potential cardiovascular adverse effects.

This is a multicenter, prospective, randomized controlled trial comparing the intraoperative arthroscopic field clarity between patients receiving epinephrine-containing irrigation and those undergoing surgery with a tourniquet.

Participants are randomized into two groups:

Epinephrine Group: Irrigation fluid consists of normal saline mixed with 1 mL of 1:1000 epinephrine per 3-liter bag. A tourniquet is placed but not inflated; it may be inflated as a rescue measure if necessary.

Tourniquet Group: Standard tourniquet application as routinely practiced.

3.2.4 Primary Efficacy Outcome

Visual field clarity (VFC) under ankle arthroscopy, assessed using a Likert-style 4-point numeric rating scale (NRS).

3.2.5 Secondary Efficacy Outcomes

Pain intensity scores at 2 and 24 hours postoperatively, measured using the Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the procedures and methods of the clinical trial
* voluntarily provide written informed consent
* Aged from 15 to 65 years old , regardless of sex
* Diagnosed with a condition requiring ankle surgery
* Be scheduled to undergo unilateral ankle arthroscopy

Exclusion Criteria:

* Patients who decline to participate in the study
* Known history of heart disease (e.g., coronary artery disease, cardiac conduction abnormalities), diabetes, or asthma
* Poorly controlled hypertension
* Age under 15 years or above 65 years old
* Intellectual disability
* Pregnant or breastfeeding women
* Known allergy to sulfites

Contraindications to ISBPB (including planned injection site infection, pre-existing neurological deficits, allergy to local anesthetics, severe chronic obstructive pulmonary disease, or contralateral phrenic nerve dysfunction)

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual field clarity (VFC) under ankle arthroscopy, assessed using a 4-point Likert-style numeric rating scale (NRS) | at 2 hours
  Scores are integers ranging from 0 to 4, with higher scores indicating clearer visual field

SECONDARY OUTCOMES:
Pain intensity at 2 and 24 hours postoperatively, assessed using the Visual Analog Scale (VAS) | at 2 and 24 hours postoperatively
  Scores range from 0 to 10, with higher scores indicating more severe pain

IPD SHARING:
Plan to Share IPD: No